CLINICAL TRIAL: NCT00345436
Title: An Exercise Intervention in Insulin-Resistant Minority Adolescents
Brief Title: Exercise in Insulin-Resistant Minority Adolescents
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906094; 06-CH-N094
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-05-11

CONDITIONS: Insulin-Resistance
Keywords: Insulin Sensitivity; Moderate intensity; Insulin Resistance; Exercise Intervention
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Insulin resistance, often accompanied by obesity, plays a major role in the development of type 2 diabetes. This phenomenon may be related with the fact that American adolescents are now becoming less physically active in early puberty, explaining the largely pubertal and post-pubertal onset of type 2 diabetes in adolescence. Although regular physical activity has been suggested to attenuate obesity and prevent type 2 diabetes in high-risk children and adolescents, the magnitude of exercise training-induced improvement in the risk factors for type 2 diabetes has been only recently studied in adults and studied very little in pediatric populations. It is clear that exercise, diet, and genetics all contribute to the development of type 2 diabetes in children. However, the few studies that have been done to dissect the relative contributions of these three risk factors have generally used only lipid profiles as the end point. There have been a number of recent advances in our understanding of the molecular basis of type 2 diabetes, particularly, with regards to insulin regulatory pathways modulated by exercise within muscle tissue.

DETAILED DESCRIPTION:
Insulin resistance, often accompanied by obesity, plays a major role in the development of type 2 diabetes. This phenomenon may be related with the fact that American adolescents are now becoming less physically active in early puberty, explaining the largely pubertal and post-pubertal onset of type 2 diabetes in adolescence. Although regular physical activity has been suggested to attenuate obesity and prevent type 2 diabetes in high-risk children and adolescents, the magnitude of exercise training-induced improvement in the risk factors for type 2 diabetes has been only recently studied in adults and studied very little in pediatric populations. It is clear that exercise, diet, and genetics all contribute to the development of type 2 diabetes in children. However, the few studies that have been done to dissect the relative contributions of these three risk factors have generally used only lipid profiles as the end point. There have been a number of recent advances in our understanding of the molecular basis of type 2 diabetes, particularly, with regards to insulin regulatory pathways modulated by exercise within muscle tissue.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be included in this study, subjects must meet the following conditions:

Sedentary (regular aerobic exercise less than or equal to 2 times/wk and less than 20 min/session): nonsmoker; impaired glucose tolerance (fasting plasma glucose greater than or equal to 100 mg/dl but less than 126 mg/dl or/and 2 hour plasma glucose greater than or equal to 140 mg/dl but less than 200 MG/dl; BMI-for-age is 95% or greater.

EXCLUSION CRITERIA:

Not pregnant; and not have any other medical condition that would preclude regular exercise.

If taking medication known to affect metabolism.

History of chronic illness known to affect metabolism.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-02-08; Study Completion 2011-05-11

CONTACTS AND LOCATIONS:
Locations (1):
- Childrens National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Arslanian S, Suprasongsin C. Differences in the in vivo insulin secretion and sensitivity of healthy black versus white adolescents. J Pediatr. 1996 Sep;129(3):440-3. doi: 10.1016/s0022-3476(96)70078-1. PMID 8804335
- [Background] Brown MD, Moore GE, Korytkowski MT, McCole SD, Hagberg JM. Improvement of insulin sensitivity by short-term exercise training in hypertensive African American women. Hypertension. 1997 Dec;30(6):1549-53. doi: 10.1161/01.hyp.30.6.1549. PMID 9403581
- [Background] Hittel DS, Kraus WE, Hoffman EP. Skeletal muscle dictates the fibrinolytic state after exercise training in overweight men with characteristics of metabolic syndrome. J Physiol. 2003 Apr 15;548(Pt 2):401-10. doi: 10.1113/jphysiol.2002.036616. Epub 2003 Feb 28. PMID 12611918
- [Derived] Many G, Hurtado ME, Tanner C, Houmard J, Gordish-Dressman H, Park JJ, Uwaifo G, Kraus W, Hagberg J, Hoffman E. Moderate-intensity aerobic training program improves insulin sensitivity and inflammatory markers in a pilot study of morbidly obese minority teens. Pediatr Exerc Sci. 2013 Feb;25(1):12-26. doi: 10.1123/pes.25.1.12. PMID 23406700